CLINICAL TRIAL: NCT04809610
Title: Effectiveness of the Internet Attachment-Based Compassion Therapy (iABCT) to Improve the Quality of Life and Well-being in a Population With Chronic Medical Illness.
Brief Title: Efficacy of Attachment-based Compassion Therapy in Population With Chronic Medical Illness (CUIDA-TEC)
Acronym: CUIDA-TEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-1564960
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-03

CONDITIONS: Chronic Medical Illness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Internet attachment-based compassion therapy (iABCT). (Experimental): The iABCT is a self-applied program based on the attachment theory and the use of compassion meditations. It is composed of 8 modules that have been reformulated to be completely self-applied and include text, images, illustrations, videos, audio with guided meditations, exercises, and homework. Downloadable PDF files will be made available so that users can review them offline. Each module has been optimized to have a duration of 60 and 90 minutes approximately. The entire intervention is estimated to be completed in eight weeks.
  Interventions: Behavioral: Internet attachment-based compassion therapy (iABCT).
- Control group: Waiting list control group. (No Intervention): Participants in this condition will be informed that they will have access to the intervention at 3 months (after the intervention group).

INTERVENTIONS:
Behavioral: Internet attachment-based compassion therapy (iABCT). — The iABCT is a self-applied program based on the attachment theory and the use of compassion meditations. It is composed of 8 modules that have been reformulated to be completely self-applied and include text, images, illustrations, videos, audio with guided meditations, exercises and homework. Downloadable PDF files will be made available so that users can review them offline. Each module has been optimized to have a duration of 60 and 90 minutes approximately. The entire intervention is estimated to be completed in eight weeks.
  Arms: Intervention group: Internet attachment-based compassion therapy (iABCT).

SUMMARY:
Compassion-Based Interventions are increasingly relevant as a potentially beneficial way to support people with chronic medical conditions and improve different outcomes related with the management of the disease. Online interventions The purpose of this study is to evaluate the effectiveness of the internet version of the attachment-based compassion therapy for improving quality of life in a population with chronic medical illness.

DETAILED DESCRIPTION:
Our participants will be randomized to one of the following two conditions: 1) the Internet version of the attachment-based compassion therapy, and 2) Waiting list (WL) control group.

The corresponding evaluations of the outcomes will be carried out at different moments of the process: baseline, and a three- and six-month follow-up.

This study will use the internet version of attachment-based compassion therapy (iABCT) for improving the quality of life in a population with chronic medical illness.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. ability to understand and read Spanish;
3. access to a computer with the Internet; and
4. fulfill criteria for diagnosis of one of the following chronic medical conditions: diabetes, inflammatory bowel disease, fibromyalgia, low-back chronic pain, migraines, and other conditions.

Exclusion Criteria:

1. Terminal disease;
2. severe psychiatric disorders comorbidities (schizophrenia, substance dependence, bipolar disorder, psychotic illness) or severe neurologic or medical condition; and
3. receiving psychological treatment or mindfulness training at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-06-22 (Estimated); Study Completion 2023-02-22 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life | Baseline (week 0), 3-month follow-up, 6-month follow-up
  EuroQol (EQ-5D; Badia et al., 1999). It is a self-report measures composed by five dimensions of functionality in daily-life and three levels of severity (1-3). A higher score in this scale indicates higher severity on the different areas of functioning in daily life.
Changes in wellbeing | Baseline (week 0), 3-month follow-up, 6-month follow-up
  Pemberton Happiness Index (PHI; Hervás and Vázquez, 2013). The scale includes eleven items related to different domains of remembered well-being (general, hedonic, eudaimonic, and social well-being) and ten items related to experienced well-being (i.e., positive and negative emotional events that possibly happened the day before); the sum of these items produces a combined well-being index that range from 0 to 10. Higher levels indicate higher levels of wellbeing.

SECONDARY OUTCOMES:
Compassion and self-compassion | Baseline (week 0), 3-month follow-up, 6-month follow-up
  Sussex-Oxford Compassion for the Self Scale (SOCS; Gu et al.,, 2020). This scale asses levels of compassion and self-compassion in a 5-point likert scale. Higher scores indicate higher levels of compassion and self-compassion.
Self-care and healthy behaviors | Baseline (week 0), 3-month follow-up, 6-month follow-up
  Mindful Self-Care Scale - Brief version (B-MSC; Cook-Cottone, 2018). It is a 24-item scale that measures the frequency of self-care behaviors. The scale addresses 6 domains of self-care: mindful relaxation, physical care, self-compassion and purpose, supportive relationships, supportive structure, and mindfulness. Higher punctuation means a higher frequency of self-care behaviors.
Specific illness interference | Baseline (week 0), 3-month follow-up, 6-month follow-up
  Specific questionnaires will be used to assess specific illness interferences for the different medical conditions included in the study: the Diabetes Distress Scale (DDS; Martin et al., 2007) for participants with type I and type II diabetes; the Roland-Morris Questionnaire (Kovacs et al., 2002) for participants with low-back chronic pain; the Revised Fibromyalgia Impact Questionnaire (FIQR; Salgueiro et al., 2013) for participants with fibromyalgia; the Migraine Disability Assessment questionnaire (MIDAS; Rodríguez-Almagro et al., 2020) for participants with migraines; and the Inflammatory Bowel Disease Questionnaire (IBDQ-32; Masachs et al., 2007) for participants with inflammatory bowel illness.
Self-criticism | Baseline (week 0), 3-month follow-up, 6-month follow-up
  Self-critical rumination Scale (SCRS; Smart et al., 2016). A 10-item questionnaire measuring self-criticism is defined as a form of negative thinking that devalues the self. It assesses thoughts that criticize the self for perceived errors, failures, weaknesses, defects, bad habits or general inadequacy. It takes into account the ruminative qualities of thought: frequency, duration, repetition, and difficulty of control. Final scores range from 10 to 40 and higher scores indicate a higher level of self-criticism.
Symptomatology | Baseline (week 0), 3-month follow-up, 6-month follow-up
  The Depression, Anxiety and Stress Scale (DASS-21; Fonseca-Pedrero et al., 2010). This scale is an abbreviated form of the DASS questionnaire containing 21 items organized in three subscales to assess anxiety, depression, and stress symptomatology. Each subscale has 7 items that range from 0 to 3 points. Higher scores indicate higher levels of symptomatology.
Attachmetn styles | Baseline (week 0), 3-month follow-up, 6-month follow-up
  The Relationships Questionnaire (RQ; Yárnoz-Yaben and Comino, 2011). This is a 4-item questionnaire designed to measure adult attachment style. The RQ consists of four paragraphs, each describing an attitude toward relationships in general. The participant rates each paragraph on a scale of 1 (does not describe me at all) to 7 (describes me exactly).
Social support | Baseline (week 0), 3-month follow-up, 6-month follow-up
  Medical Outcomes Study-Social Support Survey (MOS; Requena et al., 2007). A 20-item questionnaire that analyzes the perception of help and social support. Item 1 refers to the size of the social network and the remaining 19 items measure four dimensions of functional social support: emotional (8 items), instrumental (4 items), positive social interaction (4 items), and affective support (3 items). The items present a 5-point response scale that measures progressively (from never to always) how often each type of social support is available to the caregiver. A total score can also be obtained, where higher scores would indicate more support received.
Illness perception | Baseline (week 0), 3-month follow-up, 6-month follow-up
  Illness perception questionnaire - revised (IPQ-R; Pacheco-Huergo et al., 2012). The Illness Perception Questionnaire-Revised was designed to assess the cognitive and emotional dimensions of illness representations. The IPQ-R consists of three sections. Two scales measure the identity and causal dimensions and another section assesses the dimensions of duration (acute/chronic), cyclical course, consequences, personal control, treatment control, coherence, and emotional representations.
Client's satisfaction | 3-month follow up (only intervention group), 6-month follow-up (only WL control group)
  Expectancy and satisfaction questionnaire (adapted from Borkovec and Nau, 1972). A 6-item questionnaire that measures credibility towards treatment and patients' expectations of improvement. Higher score indicates higher levels of client credibility and expectation of improvement.
Difficulties of the compassion practice | 3-month follow-up (only intervention group), 6-month follow-up (only WL control group)
  The Compassion Practice Quality Scale (CPQS) (Navarrete et al., 2021) has been developed to assess the key aspects of compassion practices (e.g., mental imagery, sense of connection and warmth, compassionate phrases, and compassionate gestures). This self-reported questionnaire includes 10 items that participants score on a scale ranging from 0 to 100 indicating the percentage of the time that their experience reflects each statement. Higher scores indicate higher quality of practice (i.e., less practice difficulties).
Usability and client acceptance | 3-month follow-up (only intervention group), 6-month follow-up (only WL control group)
  System Usability Scale (SUS; adapted from Campos et al., 2020). The System Usability Scale (SUS) provides a reliable tool for measuring the usability of a program. It consists of a 10 item questionnaire with a 5-point likert scale. Higher scores indicate higher levels of usability and client acceptance of the program.
Semi-structured qualitative interview | 3-month follow-up (only intervention group), 6-month follow-up (only WL control group)
  An Ad-hoc instrument with open questions created to assess participants' opinions about the program and the support received. Adapted from Campos et al. 2018.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin J, Drossaert CHC, Schroevers MJ, Sanderman R, Kirby JN, Bohlmeijer ET. Compassion-based interventions for people with long-term physical conditions: a mixed methods systematic review. Psychol Health. 2021 Jan;36(1):16-42. doi: 10.1080/08870446.2019.1699090. Epub 2020 Mar 2. PMID 32116052
- [Background] Badia X, Roset M, Montserrat S, Herdman M, Segura A. [The Spanish version of EuroQol: a description and its applications. European Quality of Life scale]. Med Clin (Barc). 1999;112 Suppl 1:79-85. Spanish. PMID 10618804
- [Background] Borkovec, T. D., & Nau, S. D. (1972). Credibility of analogue therapy rationales. Journal of behavior therapy and experimental psychiatry, 3(4), 257-260.
- [Background] Campos D, Navarro-Gil M, Herrera-Mercadal P, Martinez-Garcia L, Cebolla A, Borao L, Lopez-Del-Hoyo Y, Castilla D, Del Rio E, Garcia-Campayo J, Quero S. Feasibility of the Internet Attachment-Based Compassion Therapy in the General Population: Protocol for an Open-Label Uncontrolled Pilot Trial. JMIR Res Protoc. 2020 Aug 14;9(8):e16717. doi: 10.2196/16717. PMID 32384051
- [Background] Cook-Cottone, C. P., & Guyker, W. M. (2018). The development and validation of the Mindful Self-Care Scale (MSCS): An assessment of practices that support positive embodiment. Mindfulness, 9(1), 161-175.
- [Background] Del Re AC, Fluckiger C, Goldberg SB, Hoyt WT. Monitoring mindfulness practice quality: an important consideration in mindfulness practice. Psychother Res. 2013;23(1):54-66. doi: 10.1080/10503307.2012.729275. Epub 2012 Oct 9. PMID 23046287
- [Background] Fonseca-Pedrero, E., Paino, M., Lemos-Giráldez, S., & Muñiz, J. (2010). Propiedades psicométricas de la depression anxiety and stress scales-21 (DASS-21) en universitarios españoles. Ansiedad y Estrés, 16.
- [Background] Finlay-Jones A, Boyes M, Perry Y, Sirois F, Lee R, Rees C. Online self-compassion training to improve the wellbeing of youth with chronic medical conditions: protocol for a randomised control trial. BMC Public Health. 2020 Jan 28;20(1):106. doi: 10.1186/s12889-020-8226-7. PMID 31992269
- [Background] Gu J, Baer R, Cavanagh K, Kuyken W, Strauss C. Development and Psychometric Properties of the Sussex-Oxford Compassion Scales (SOCS). Assessment. 2020 Jan;27(1):3-20. doi: 10.1177/1073191119860911. Epub 2019 Jul 29. PMID 31353931
- [Background] Hervas G, Vazquez C. Construction and validation of a measure of integrative well-being in seven languages: the Pemberton Happiness Index. Health Qual Life Outcomes. 2013 Apr 22;11:66. doi: 10.1186/1477-7525-11-66. PMID 23607679
- [Background] Irani E, Niyomyart A, Hickman RL Jr. Systematic Review of Technology-Based Interventions Targeting Chronically Ill Adults and Their Caregivers. West J Nurs Res. 2020 Nov;42(11):974-992. doi: 10.1177/0193945919897011. Epub 2020 Jan 16. PMID 31941418
- [Background] Pacheco-Huergo V, Viladrich C, Pujol-Ribera E, Cabezas-Pena C, Nunez M, Roura-Olmeda P, Amado-Guirado E, Nunez E, Del Val JL; en representacion del Grupo IPQ-R. [Perception in chronic illnesses: linguistic validation of the revised Illness Perception Questionnaire and the Brief Illness Perception Questionnaire for a Spanish population]. Aten Primaria. 2012 May;44(5):280-7. doi: 10.1016/j.aprim.2010.11.022. Epub 2011 Sep 28. Spanish. PMID 21955598
- [Background] Costa Requena G, Salamero M, Gil F. [Validity of the questionnaire MOS-SSS of social support in neoplastic patients]. Med Clin (Barc). 2007 May 12;128(18):687-91. doi: 10.1157/13102357. Spanish. PMID 17540143
- [Background] Rogers MA, Lemmen K, Kramer R, Mann J, Chopra V. Internet-Delivered Health Interventions That Work: Systematic Review of Meta-Analyses and Evaluation of Website Availability. J Med Internet Res. 2017 Mar 24;19(3):e90. doi: 10.2196/jmir.7111. PMID 28341617
- [Background] Sirois, F. M., Molnar, D. S., & Hirsch, J. K. (2015). Self-compassion, stress, and coping in the context of chronic illness. Self and Identity, 14(3), 334-347.
- [Background] Smart LM, Peters JR, Baer RA. Development and Validation of a Measure of Self-Critical Rumination. Assessment. 2016 Jun;23(3):321-32. doi: 10.1177/1073191115573300. Epub 2015 Feb 23. PMID 25712674
- [Background] Yárnoz-Yaben, S., & Comino, P. (2011). Evaluación del apego adulto: análisis de la convergencia entre diferentes instrumentos. Acción psicológica, 8(2), 67-85.
- [Derived] Martinez-Sanchis M, Vara MD, Herrero R, Campos D, Garcia-Campayo J, Banos RM. Effectiveness of the Internet Attachment-Based Compassion Therapy (iABCT) to improve the quality of life and well-being in a population with chronic medical illness: A study protocol of a randomized controlled trial (SPIRIT compliant). PLoS One. 2022 Dec 27;17(12):e0278462. doi: 10.1371/journal.pone.0278462. eCollection 2022. PMID 36574408